CLINICAL TRIAL: NCT02492711
Title: A Phase 3, Randomized Study of Margetuximab Plus Chemotherapy vs Trastuzumab Plus Chemotherapy in the Treatment of Patients With HER2+ Metastatic Breast Cancer Who Have Received Prior Anti-HER2 Therapies and Require Systemic Treatment
Brief Title: Margetuximab Plus Chemotherapy vs Trastuzumab Plus Chemotherapy in the Treatment of HER2+ Metastatic Breast Cancer
Acronym: SOPHIA
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: MacroGenics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CP-MGAH22-04
Record Dates: First submitted 2015-07-06; First posted 2015-07-09 (Estimated); Results first posted 2022-11-23 (Actual); Last update posted 2025-03-17 (Actual); Status verified 2025-02

CONDITIONS: HER-2 Positive Breast Cancer; Metastatic Neoplasm
MeSH Terms: conditions — Neoplasm Metastasis | interventions — margetuximab; Trastuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Margetuximab plus chemotherapy (Experimental): Margetuximab 15 mg/kg every 21 days
  Interventions: Biological: Margetuximab; Drug: Physician's choice of chemotherapy.
- Trastuzumab plus chemotherapy (Active Comparator): Trastuzumab 8 mg/kg loading dose, then 6 mg/kg every 21 days
  Interventions: Biological: Trastuzumab; Drug: Physician's choice of chemotherapy.
- Margetuximab Infusion Sub-study (Experimental): Margetuximab 15 mg/kg every 21 days (with or without chemotherapy), studying a shorter duration of infusion beginning in Cycle 2.
  Interventions: Biological: Margetuximab; Drug: Physician's choice of chemotherapy.

INTERVENTIONS:
Biological: Margetuximab — 15 mg/kg via IV (intravenous) infusion on day 1 of each 21 day cycle,
  Other Names: MGAH22; Margenza®
  Arms: Margetuximab Infusion Sub-study; Margetuximab plus chemotherapy
Biological: Trastuzumab — 8 mg/kg via IV (intravenous) infusion for the first dose and 6 mg/kg for all subsequent doses via IV infusion on day 1 of each 21 day cycle
  Other Names: Herceptin®
  Arms: Trastuzumab plus chemotherapy
Drug: Physician's choice of chemotherapy. — Capecitabine (Xeloda®):1000 mg/m2 BID for 14 days in a 21-day cycle, or Eribulin (Halaven®): 1.4 mg/m2 on days 1 and 8 of a 21-day cycle, or Gemcitabine (Gemzar®): 1000 mg/m2 on days 1 and 8 of a 21-day cycle, or Vinorelbine (Navelbine®): 25-30 mg/m2 on days 1 and 8 of a 21-day cycle

SUMMARY:
The purpose of this study is to determine whether patients with metastatic breast cancer treated with margetuximab plus chemotherapy have longer progression free survival (PFS) and overall survival (OS) than patients treated with trastuzumab plus chemotherapy.

A non-randomized sub-study cohort of approximately 88 patients will be enrolled to evaluate the safety of a reduced margetuximab infusion rate in patients receiving margetuximab either as monotherapy or in combination with chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Histologically-proven metastatic or locally-advanced relapsed/refractory HER2+ breast cancer based on the most recently available tumor biopsy collected from the patient. Tumors may be estrogen receptor (ER)/progesterone receptor (PgR) positive or negative.
* Have received at least 2 prior lines of anti-HER2 directed therapy in the metastatic setting, or in case of having received (neo)adjuvant pertuzumab, at least 1 prior line of anti-HER2 directed therapy in the metastatic setting. In either case, patients must have received prior treatment with pertuzumab, in the (neo)adjuvant or metastatic setting. Prior radiotherapy, hormonal therapies, and other anti-HER2 therapies are allowed.
* Prior treatment with at least one, and no more than three, lines of therapy overall in the metastatic setting. Patients must have progressed on or following, the most recent line of therapy.
* Resolution of all chemotherapy or radiation-related toxicities to ≤ Grade 1
* Life expectancy ≥ 12 weeks
* Acceptable laboratory parameters
* Women of childbearing potential must have negative pregnancy test performed within 14 days of randomization and on the first day of treatment. All subjects must agree to use an effective form of contraception for the duration of study treatment and for 7 months after the last dose of study drug.

Infusion sub-study prior therapy requirements: Same as above, except:

* Must have received 4 or more prior lines or therapy in the metastatic setting
* Must have received prior trastuzumab, pertuzumab, and T-DM1

Exclusion Criteria:

* Known, untreated brain metastasis. Patients with signs or symptoms of brain metastasis must have a CT or MRI performed within 4 weeks prior to randomization to specifically exclude the presence of radiographically-detected brain metastases
* History of uncontrolled seizures within 6 months of randomization
* History of prior allogeneic bone marrow, stem-cell, or solid organ transplantation
* History of clinically significant cardiovascular disease
* Clinically-significant pulmonary compromise, including a requirement for supplemental oxygen use to maintain adequate oxygenation
* Any condition that would be a contraindication to receiving trastuzumab as described in the approved local label or a condition that would prevent treatment with the physician's choice of chemotherapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 624 (Actual)
Dates: Start 2015-08-24 (Actual); Primary Completion 2021-08-11 (Actual); Study Completion 2022-06-14 (Actual)

CONTACTS AND LOCATIONS:
Locations (167):
- United States (62):
  - Ironwood Cancer & Research Center, Chandler, Arizona
  - Banner MD Anderson Cancer Center, Gilbert, Arizona
  - Western Regional Medical Center, Inc., Goodyear, Arizona
  - East Valley Hematology And Oncology, Burbank, California
  - UCLA Hematology Oncology Santa Monica, Los Angeles, California
  - UC Davis Comprehensive Cancer Center, Sacramento, California
  - Sharp Memorial Hospital, San Diego, California
  - University of California, San Francisco Helen Diller Family Comprehensive Cancer Center, San Francisco, California
  - Kaiser Permenente Medical Center, Vallejo, California
  - Poudre Valley Health Care, Inc., Fort Collins, Colorado
  - MedStar Washington Hospital Center, Washington D.C., District of Columbia
  - Florida Cancer Specialists, Fort Myers, Florida
  - Memorial Cancer Institute at Memorial Regional Hospital, Hollywood, Florida
  - Mount Sinai Comprehensive Cancer Center, Miami Beach, Florida
  - Florida Cancer Specialists, New Port Richey, Florida
  - Orlndo Health Cancer Center, Orlando, Florida
  - Hem-Onc Associates, Port Saint Lucie, Florida
  - Palm Beach Cancer Center, West Palm Beach, Florida
  - Piedmont Cancer Institute, P.C., Atlanta, Georgia
  - Northwest Georgia Oncology Centers, PC, Marietta, Georgia
  - CTCA - Southeastern Regional Medical Center, Newnan, Georgia
  - Kaiser Permanente Hawaii Moanalua Medical Center, Honolulu, Hawaii
  - Northwestern University Feinberg School of Medicine, Chicago, Illinois
  - Rush University Medical Center, Chicago, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - CTCA - Midwestern Regional Medical Center, Zion, Illinois
  - Indiana University Health Goshen Center for Cancer Care, Goshen, Indiana
  - ARH Cancer Clinic, Hazard, Kentucky
  - St. Joseph's Hospital, Lexington, Kentucky
  - Touro Infirmary Hospital, New Orleans, Louisiana
  - New England Cancer Specialists, Scarborough, Maine
  - Mercy Medical Center, Baltimore, Maryland
  - Tufts-NEMC Cancer Center, Boston, Massachusetts
  - Forrest General Hospital, Hattiesburg, Mississippi
  - Saint Luke's Cancer Specialists, Kansas City, Missouri
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - Dartmouth-Hitchcock - Norris C, Lebanon, New Hampshire
  - New Jersey Hematology Oncology Associates, Brick, New Jersey
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Saint Barnabas Medical Center - The Cancer Center, Livingston, New Jersey
  - New Mexico Cancer Care Alliance (NMCCA), Albuquerque, New Mexico
  - Queens Hospital Center, Jamaica, New York
  - ProHEALTH CARE Associates, LLP, Lake Success, New York
  - New York University Clinical Cancer Center, New York, New York
  - Wake Forest University Baptist Medical Center (WFUBMC), Winston-Salem, North Carolina
  - Mercy Physicians Of Oklahoma, Oklahoma City, Oklahoma
  - Pinnacle Health Cancer Institute, Harrisburg, Pennsylvania
  - Monongahela Valley Hospital, Monongahela, Pennsylvania
  - CTCA - Eastern Regional Medical Center, Inc., Philadelphia, Pennsylvania
  - Guthrie Medical Group, PC, Sayre, Pennsylvania
  - Tennessee Oncology, PLLC, Chattanooga, Tennessee
  - The Sarah Cannon Research Institute, Nashville, Tennessee
  - Austin Cancer Center, Austin, Texas
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - The Center for Cancer and Blood Disorders, Fort Worth, Texas
  - Utah Cancer Specialists, Salt Lake City, Utah
  - University of Virginia Cancer Center, Charlottesville, Virginia
  - Inova Schar Cancer Institute, Fairfax, Virginia
  - Fort Belvoir Community Hospital, Fort Belvoir, Virginia
  - Swedish Cancer Institute/ Swedish Health Services, Seattle, Washington
  - University of Washington/ Seattle Cancer Care Alliance, Seattle, Washington
  - Cancer Care Northwest, PS, Spokane, Washington
- Medizinische Universität Innsbruck, Innsbruck, Tyrol, Austria
- Belgium (12):
  - UZ Antwerpen, Edegem, Antwerpen
  - GZA Ziekenhuizen - Campus Sint-Augustinus, Wilrijk, Antwerpen
  - Clinique Saint-Pierre Ottignies, Ottignies, Brabant Wallon
  - UZ Brussel - Campus Jette, Brussels, Brussels Capital
  - Cliniques universitaires Saint-Luc, Brussels, Brussels Capital
  - Jessa Ziekenhuis - Campus Virga Jesse, Hasselt, Limburg
  - AZ Nikolaas - Campus Sint-Niklaas Moerland, Sint-Niklaas, Oost-Vlaanderen
  - AZ Sint-Jan Brugge - Oostende - Campus Sint-Jan, Bruges, West-Vlaanderen
  - AZ Groeninge - Campus Loofstraat, Kortrijk, West-Vlaanderen
  - AZ Damiaan, Ostend, West-Vlaanderen
  - Chc - Clinique Saint-Joseph, Liège
  - Clinique Sainte Elisabeth, Namur
- Canada (2):
  - Dr. Leon Richard Oncology Centre, Moncton, New Brunswick
  - Lakeridge Health Oshawa, Oshawa, Ontario
- Czechia (3):
  - Masarykuv onkologicky ustav, Brno, Brno-město
  - Fakultni nemocnice Olomouc, Olomouc
  - Fakultni nemocnice v Motole, Prague
- Denmark (4):
  - Aarhus Universitetshospital, Aarhus C, Central Jutland
  - Regionshospitalet Herning (Herning Centralsygehus), Herning, Central Jutland
  - Vejle Sygehus, Vejle, Region Syddanmark
  - Næstved Sygehus, Aarhus N, Zeeland
- Finland (2):
  - Tampere University Hospital, Tampere, Etelä-Suomen Lääni
  - Helsinki University Central Hospital (HUCH) - Meilahden Sair, Helsinki, Länsi-Suomen Lääni
- France (8):
  - Center de Lutte Contre le Cancer (CLCC), Nice, Alpes-Martitimes
  - Centre Léon Bérard, Lyon, Auvergne-Rhône-Alpes
  - Center de Lutte Contre le Cancer (CLCC), Caen, Calvados
  - Centre Georges-François Lecler, Dijon, Côte-d'Or
  - Centre de Lutte Contre le Cancer (CLCC) - Institut de Cancer, Saint-Herblain, Loire-Atlantique
  - Centre Jean Perrin, Clermont-Ferrand, Puy-de-Dôme
  - Institut Curie, Paris, Île-de-France Region
  - Institut Curie - Hôpital René Huguenin, Saint-Cloud, Île-de-France Region
- Germany (8):
  - Universitaetsklinikum Tuebingen, Tübingen, Baden-Wurttemberg
  - Universitätsklinikum Erlangen, Erlangen, Bavaria
  - Praxis für Frauenheilkunde Anita, München, Bavaria
  - Marien Hospital Düsseldorf, Düsseldorf, Nordhein-Westfalen
  - Universitaetsklinikum Essen - Klinik fuer Frauenheilkunde, Essen, North Rhine-Westphalia
  - Marien Hospital, Witten, North Rhine-Westphalia
  - Medizinische Fakultät Carl Gustav Carus, Dresden, Saxony
  - Universtatsklinikum Heidelberg Nationales, Heidelberg
- Israel (8):
  - Meir Medical Center, Kfar Saba, Central District
  - Rabin Medical Center - Beilinson Hospital, Petah Tikva, Central District
  - The Chaim Sheba Medical Center - Insititute of Oncology, Ramat Gan, Central District
  - Kaplan Medical Center, Rehovot, Central District
  - Hadassah Medical Organisation, Hadassah Medical Center, Ein-Karem, Jerusalem, Jerusalem
  - Soroka Medical Center [Oncology], Beersheba, Southern District
  - Clalit Health Services - Lin Medical Center, Haifa
  - Tel Aviv Sourasky Medical Center, Tel Aviv
- Italy (23):
  - PO Garibaldi-Nesima, ARNAS Garibaldi, Catania, Cantania
  - Irccs Irst, Meldola, Forli
  - Istituto di Candiolo, IRCCS, Candiolo, Torino
  - Azienda Ospedaliero Universitaria Senese Universita degli St, Siena, Tuscany
  - Ospedale Umberto I, AOU Ospedali Riuniti Umberto I - GM.Lanc, Ancona
  - AO G.Rummo, Benevento
  - ASST Papa Giovanni XXIII - Oncologia-Bergamo, Bergamo
  - PO di Cremona, ASST di Cremona - Patologia Mammaria e Breast Unit - Cremona, Cremona
  - Arcispedale S.Anna, AOU di Ferrara, Ferrara
  - E.O. Ospedali Galliera, Genova
  - PO A.Manzoni di Lecco, ASST Lecco - Oncologia Medica - Lecco, Lecco
  - Azienda Ospedaliera Fatebenefratelli e Oftalmico, Milan
  - Istituto Europeo di Oncologia Via Ripamonti, Milan
  - AOU Policlinico di Modena, Modena
  - Fondazione Pascale, IRCCS Istituto Nazionale dei Tumori, Napoli
  - AOU di Parma, Parma
  - IRCCS Policlinico San Matteo, Pavia
  - IRCSS Fodazione Salvatore Maugeri, Pavia
  - SO S.Chiara, AOU Pisana, Pisa
  - Nuovo ospedale di Prato, Prato
  - PU Campus Bio-medico di Roma, Roma
  - AO S.Andrea, Università degli Studi di Roma La Sapienza, Roma
  - Ospedale Belcolle Viterbo, Viterbo
- Netherlands (2):
  - Maastricht University Medical Centre, Maastricht, Limburg
  - Haga Ziekenhuis, loc. Leyenburg, The Hague, South Holland
- Poland (3):
  - MAGODENT Sp. z o.o., Warsaw, Masovian Voivodeship
  - Mazowiecki Szpital Onkologiczny, Wieliszew, Masovian Voivodeship
  - Centrum Onkologii Ziemi Lubelskiej im. Sw. Jana z Dukli, Lublin
- Portugal (3):
  - Centro Clínico Champalimaud/Fundação Champalimaud, Lisbon, Lisbon District
  - H. Santa Maria - Centro Hospitalar Lisboa Norte, Lisbon
  - Instituto Português Oncologia Francisco Gentil do Porto, Porto
- Fundacion de Investigacion de Diego, San Juan, Puerto Rico
- South Korea (4):
  - Seoul National University Hospital, Seoul, Seoul Teugbyeolsi
  - Severance Hospital, Yonsei University Health System, Seoul, Seoul Teugbyeolsi
  - Asan Medical Center, Seoul, Seoul Teugbyeolsi
  - Samsung Medical Center, Seoul, Seoul Teugbyeolsi
- Spain (16):
  - H.U.V. del Rocío, Seville, Andalusia
  - Institut Català d'Oncologia-Hospital Germans Trias i Pujol, Badalona, Barcelona
  - Hospital Universitari Parc Taulí, Sabadell, Barcelona
  - Hospital del Mar, Barcelona, Catalonia
  - H.C.U. Valencia, Valencia, Comunidad
  - Hospital de Navarra, Pamplona, Navarre
  - H.U. Sant Joan de Reus, Reus, Tarragona
  - Hospital Ntra. Sra. de Sonsoles, Ávila
  - Hospital Universitario Vall d'Hebron, Barcelona
  - H. San Pedro de Alcántara, Cáceres
  - H.U. Arnau de Vilanova, Lleida
  - M.D. Anderson Cancer Center Madrid, Madrid
  - Hospital Universitario Ramón y Cajal, Madrid
  - Hospital Universitario Clínico San Carlos, Madrid
  - Fundación Instituto Valenciano de Oncología, Valencia
  - Hospital Universitari I Politecnic La Fe, Valencia
- United Kingdom (5):
  - Guys and St Thomas Hospital, London, City of London
  - Castle Hill Hospital (Hull), Hull, East Riding Of Yorkshire
  - Kent Oncology Centre, Maidstone Hospital, Maidstone, Kent
  - Royal Preston Hospital, Fulwood, Lancashire
  - South Tees Hospitals NHS Foundation Trust, Middlesbrough

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Rugo HS, Im SA, Cardoso F, Cortes J, Curigliano G, Musolino A, Pegram MD, Bachelot T, Wright GS, Saura C, Escriva-de-Romani S, De Laurentiis M, Schwartz GN, Pluard TJ, Ricci F, Gwin WR 3rd, Levy C, Brown-Glaberman U, Ferrero JM, de Boer M, Kim SB, Petrakova K, Yardley DA, Freedman O, Jakobsen EH, Gal-Yam EN, Yerushalmi R, Fasching PA, Kaufman PA, Ashley EJ, Perez-Olle R, Hong S, Rosales MK, Gradishar WJ; SOPHIA Study Group. Margetuximab Versus Trastuzumab in Patients With Previously Treated HER2-Positive Advanced Breast Cancer (SOPHIA): Final Overall Survival Results From a Randomized Phase 3 Trial. J Clin Oncol. 2023 Jan 10;41(2):198-205. doi: 10.1200/JCO.21.02937. Epub 2022 Nov 4. PMID 36332179
- [Derived] Rugo HS, Im SA, Cardoso F, Cortes J, Curigliano G, Musolino A, Pegram MD, Wright GS, Saura C, Escriva-de-Romani S, De Laurentiis M, Levy C, Brown-Glaberman U, Ferrero JM, de Boer M, Kim SB, Petrakova K, Yardley DA, Freedman O, Jakobsen EH, Kaufman B, Yerushalmi R, Fasching PA, Nordstrom JL, Bonvini E, Koenig S, Edlich S, Hong S, Rock EP, Gradishar WJ; SOPHIA Study Group. Efficacy of Margetuximab vs Trastuzumab in Patients With Pretreated ERBB2-Positive Advanced Breast Cancer: A Phase 3 Randomized Clinical Trial. JAMA Oncol. 2021 Apr 1;7(4):573-584. doi: 10.1001/jamaoncol.2020.7932. PMID 33480963

RESULTS

PARTICIPANT FLOW:
Groups:
- Margetuximab Plus Chemotherapy: Margetuximab 15 mg/kg administered every 21 days with physician's choice of 1 of 4 backbone chemotherapy regimens.
- Trastuzumab Plus Chemotherapy: Trastuzumab administered every 21 days with physician's choice of 1 of 4 backbone chemotherapy regimens.
- Margetuximab Infusion Substudy: Margetuximab with or without chemotherapy administered as a 120 minute first infusion in Cycle 1 followed by 60-minute or 30-minute infusion in Cycle 2.
Period: Overall Study
Arm/Group | Margetuximab Plus Chemotherapy | Trastuzumab Plus Chemotherapy | Margetuximab Infusion Substudy
Started | 266 | 270 | 88
Intent-to-treat (ITT) Population | 266 | 270 | 88
Safety Population | 264 | 266 | 88
Completed | 230 | 230 | 75
Not Completed | 36 | 40 | 13
Not completed — Adverse Event | 9 | 9 | 2
Not completed — Death | 3 | 3 | 0
Not completed — Withdrawal by Subject | 10 | 16 | 5
Not completed — Physician Decision | 10 | 6 | 4
Not completed — Lost to Follow-up | 0 | 0 | 1
Not completed — study treatment delay | 2 | 1 | 0
Not completed — change in chemotherapy | 0 | 1 | 0
Not completed — never treated | 2 | 4 | 0
Not completed — Other | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Margetuximab Infusion Substudy: Margetuximab with or without chemotherapy
- Total: Total of all reporting groups
Arm/Group | Margetuximab Plus Chemotherapy | Trastuzumab Plus Chemotherapy | Margetuximab Infusion Substudy | Total
Number analyzed (Participants) | 266 | 270 | 88 | 624
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.4 (11.4) | 55.7 (11.5) | 54.5 (12.5) | 55.1 (11.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 266 | 267 | 87 | 620
  Male | 0 | 3 | 1 | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 16 | 30 | 7 | 53
  Not Hispanic or Latino | 217 | 214 | 75 | 506
  Unknown or Not Reported | 33 | 26 | 6 | 65
Race (NIH/OMB) [Count of Participants; unit: Participants]
  other: American Indian or Alaska Native | 0 | 0 | 0 | 0
  other: Asian | 20 | 14 | 9 | 43
  other: Native Hawaiian or Other Pacific Islander | 1 | 2 | 0 | 3
  other: Black or African American | 16 | 12 | 8 | 36
  other: White | 205 | 222 | 62 | 489
  other: More than one race | 0 | 0 | 9 | 9
  other: Unknown or Not Reported | 24 | 20 | 0 | 44
Region of Enrollment [Number; unit: participants]
  Belgium | 12 | 13 | 6 | 31
  Canada | 4 | 6 | 2 | 12
  Czechia | 4 | 8 | 0 | 12
  France | 22 | 13 | 5 | 40
  Israel | 12 | 20 | 9 | 41
  Italy | 41 | 33 | 15 | 89
  South Korea | 16 | 9 | 6 | 31
  Portugal | 5 | 6 | 2 | 13
  Puerto Rico | 1 | 1 | 2 | 4
  United States | 81 | 96 | 41 | 218
  Austria | 3 | 1 | 0 | 4
  Finland | 3 | 1 | 0 | 4
  Denmark | 9 | 7 | 0 | 16
  Germany | 10 | 7 | 0 | 17
  Netherlands | 3 | 4 | 0 | 7
  Poland | 4 | 6 | 0 | 10
  Spain | 27 | 34 | 0 | 61
  United Kingdom | 9 | 5 | 0 | 14

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival (PFS) as Determined by Independent Radiological Review.
Description: PFS is measured from the time of randomization until first documented disease progression or death from any cause, whichever is first.
Time Frame: Tumor assessments are conducted every 6 weeks for the first 24 weeks and then every 24 weeks until progression of cancer, average 5 months.
Population: The PFS outcome measure is calculated only for the randomized study efficacy population. The 88 participants in the sub-study were not part of the efficacy population
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Margetuximab Infusion Substudy: Margetuximab with or without chemotherap...
Arm/Group | Margetuximab Plus Chemotherapy | Trastuzumab Plus Chemotherapy | Margetuximab Infusion Substudy
Number analyzed (Participants) | 266 | 270 | 0
months | 5.8 [5.52 to 6.97] | 4.9 [4.17 to 5.59] |
Statistical Analysis 1: Comparison: Margetuximab Plus Chemotherapy vs Trastuzumab Plus Chemotherapy; Test type: Superiority; p = 0.0334, Log Rank; Stratified Log-Rank Test; Hazard Ratio (HR) = 0.76, 95% CI 2-sided [0.593 to 0.979] — Stratified Cox Proportional Model

2. Primary Outcome: Overall Survival (OS) Defined as the Number of Days From Randomization to the Date of Death (From Any Cause).
Description: Overall survival is the time from randomization until death from any cause
Time Frame: Throughout the study, average 21 months
Population: The OS outcome measure is calculated only for the randomized study efficacy population. The 88 participants in the sub-study were not part of the efficacy population
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Margetuximab Plus Chemotherapy | Trastuzumab Plus Chemotherapy | Margetuximab Infusion Substudy
Number analyzed (Participants) | 266 | 270 | 0
months | 21.6 [0.66 to 61.44] | 21.9 [0.07 to 64.53] |
Statistical Analysis 1: Comparison: Margetuximab Plus Chemotherapy vs Trastuzumab Plus Chemotherapy; Test type: Superiority; p = 0.6204, Log Rank; Stratified Log-Rank Test; Hazard Ratio (HR) = 0.950, 95% CI 2-sided [0.774 to 1.165] — Stratified Cox Proportional Model

3. Primary Outcome: Number of Patients With Grade 3 or Higher Infusion Related Reactions
Description: Incidence of Grade 3 or higher infusion-related reactions for patients receiving 60-minute or 30-minute infusions of margetuximab in Cycle 2 of treatment
Time Frame: 22 days
Population: Only patients in the infusion substudy are included in this outcome measure.
Measure: Count of Participants; unit: Participants
Groups:
- Margetuximab Stage A1: Margetuximab administered as a 120 minute first infusion in Cycle 1 followed by 60 minute infusion in Cycle 2.
- Margetuximab Stage A2; Margetuximab Stage B: Margetuximab administered as a 120 minute first infusion in Cycle 1 followed by 30 minute infusion in Cycle 2.
Arm/Group | Margetuximab Plus Chemotherapy | Trastuzumab Plus Chemotherapy | Margetuximab Stage A1 | Margetuximab Stage A2 | Margetuximab Stage B
Number analyzed (Participants) | 0 | 0 | 8 | 9 | 71
Participants |  |  | 0 | 0 | 0

4. Secondary Outcome: To Evaluate Progression-free Survival (PFS), as Assessed by Study Investigators.
Time Frame: Tumor assessments are conducted every 6 weeks for the first 24 weeks and then every 24 weeks until progression of cancer, up to 6.5 years.
Population: Analysis population consisted of all patient who had investigator-assessed responses to treatment as of the interim analysis. The outcome measure is calculated only for the randomized study population. The 88 participants in the sub-study were not part of the efficacy population.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Margetuximab Plus Chemotherapy | Trastuzumab Plus Chemotherapy | Margetuximab Infusion Substudy
Number analyzed (Participants) | 160 | 177 | 0
months | 5.6 [5.06 to 6.67] | 4.2 [3.98 to 5.39] |
Statistical Analysis 1: Comparison: Margetuximab Plus Chemotherapy vs Trastuzumab Plus Chemotherapy; Test type: Superiority; p = 0.0014, Log Rank; Stratified Log-Rank Test; Hazard Ratio (HR) = 0.70, 95% CI 2-sided [0.556 to 0.870] — Stratified Cox Proportional Model

5. Secondary Outcome: To Evaluate the Objective Response Rate (ORR) as Determined by Independent Radiological Review.
Description: Objective response rate includes all patients with either a complete response (CR) or a partial response (PR) to study treatment
Time Frame: as for outcome 4
Population: Tumor response was assessed for patients with measurable disease at baseline. The cutoff data for analysis corresponds with the completion of enrollment. Detection of ORR requires at least 12 weeks, so the ORR may be underestimated. Outcome measure is calculated only for the randomized study population. The 88 participants in the sub-study were not part of the efficacy population.
Measure: Count of Participants; unit: Participants
Arm/Group | Margetuximab Plus Chemotherapy | Trastuzumab Plus Chemotherapy | Margetuximab Infusion Substudy
Number analyzed (Participants) | 262 | 262 | 0
Participants
  CR | 7 | 4 |
  PR | 51 | 38 |
  No response, progressive disease, not evaluable or not available | 204 | 220 |

6. Secondary Outcome: Infusion Rate Sub-study All Safety
Description: Incidence of all grades of infusion-related reactions
Time Frame: Throughout the study, average duration 6 months
Population: Only patients in the infusion substudy were evaluated for this outcome measure
Measure: Number; unit: participants
Arm/Group | Margetuximab Plus Chemotherapy | Trastuzumab Plus Chemotherapy | Margetuximab Stage A1 | Margetuximab Stage A2 | Margetuximab Stage B
Number analyzed (Participants) | 0 | 0 | 8 | 9 | 71
participants
  Infusion related reaction Cycle 1 |  |  | 1 | 1 | 16
  Infusion related reaction Cycle 2 or higher |  |  | 0 | 0 | 2
  No infusion related reaction |  |  | 7 | 8 | 55

ADVERSE EVENTS:
Time Frame: AEs were collected from the time of first dose through 30 days after the last dose, average 6 months. All-cause mortality was collected from the first dose until the primary completion date, average 2 years.
Description: AEs are based on physical exam, patient reports, and significant abnormal laboratory values.
  AEs were not collected in survival follow up. Only SAEs were collected in survival follow up if related to study treatment.
  Only patients who received study treatments were assessed for safety. All patients in the ITT population were assessed for all-cause mortality.
  Progression of cancer causing hospitalization or death is not considered an SAE, unless considered drug-related by the investigator.
Groups:
- Margetuximab Plus Chemotherapy; Trastuzumab Plus Chemotherapy: Trastuzumab administered every 21 days with physician's choice of 1 of 4 backbone chemotherapy regimens.
Arm/Group | Margetuximab Plus Chemotherapy | Trastuzumab Plus Chemotherapy | Margetuximab Infusion Substudy
All-Cause Mortality (participants affected / at risk) | 194/266 | 191/270 | 56/88
Serious Adverse Events (participants affected / at risk) | 47/264 | 51/266 | 17/88
Other Adverse Events (participants affected / at risk) | 213/264 | 210/266 | 68/88
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Margetuximab Plus Chemotherapy (N=264) | Trastuzumab Plus Chemotherapy (N=266) | Margetuximab Infusion Substudy (N=88)
Febrile neutropenia (Blood and lymphatic system disorders) | 4 | 10 | 0
Anaemia (Blood and lymphatic system disorders) | 2 | 2 | 1
Neutropenia (Blood and lymphatic system disorders) | 4 | 1 | 0
Acute myocardial infarction (Cardiac disorders) | 1 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 1 | 0
Cardiac failure (Cardiac disorders) | 1 | 0 | 0
Ventricular tachycardia (Cardiac disorders) | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 1 | 2
Constipation (Gastrointestinal disorders) | 1 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 1
Vomiting (Gastrointestinal disorders) | 1 | 0 | 1
Colitis (Gastrointestinal disorders) | 1 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 1
Gastrointestinal toxicity (Gastrointestinal disorders) | 0 | 1 | 0
Impaired gastric emptying (Gastrointestinal disorders) | 1 | 0 | 0
Intestinal obstruction (Gastrointestinal disorders) | 0 | 1 | 0
Irritable bowel syndrome (Gastrointestinal disorders) | 1 | 0 | 0
Large intestine perforation (Gastrointestinal disorders) | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 0 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 1
Pyrexia (General disorders) | 2 | 3 | 1
General physical health deterioration (General disorders) | 0 | 1 | 1
Malaise (General disorders) | 1 | 1 | 0
Asthenia (General disorders) | 0 | 1 | 0
Chills (General disorders) | 0 | 1 | 0
Death (General disorders) | 1 | 0 | 0
Infusion site extravasation (General disorders) | 1 | 0 | 0
Non-cardiac chest pain (General disorders) | 0 | 1 | 0
Pain (General disorders) | 0 | 0 | 1
Allergic oedema (Immune system disorders) | 1 | 0 | 0
Pneumonia (Infections and infestations) | 4 | 8 | 1
Cellulitis (Infections and infestations) | 1 | 3 | 0
Urinary tract infection (Infections and infestations) | 2 | 2 | 0
Influenza (Infections and infestations) | 1 | 2 | 0
Breast cellulitis (Infections and infestations) | 0 | 2 | 0
Bronchitis (Infections and infestations) | 0 | 1 | 1
Septic shock (Infections and infestations) | 1 | 0 | 1
Acinetobacter infection (Infections and infestations) | 0 | 1 | 0
Breast abscess (Infections and infestations) | 0 | 1 | 0
Catheter site infection (Infections and infestations) | 0 | 0 | 1
Clostridium difficile infection (Infections and infestations) | 0 | 1 | 0
Corona virus infection (Infections and infestations) | 1 | 0 | 0
Device related infection (Infections and infestations) | 1 | 0 | 0
Device related sepsis (Infections and infestations) | 0 | 1 | 0
Gastroenteritis (Infections and infestations) | 0 | 1 | 0
Gastroenteritis viral (Infections and infestations) | 0 | 1 | 0
Infected bite (Infections and infestations) | 0 | 1 | 0
Infection (Infections and infestations) | 1 | 0 | 0
Lung infection (Infections and infestations) | 0 | 1 | 0
Mastitis (Infections and infestations) | 1 | 0 | 0
Mastoiditis (Infections and infestations) | 1 | 0 | 0
Periorbital cellulitis (Infections and infestations) | 1 | 0 | 0
Pseudomonal sepsis (Infections and infestations) | 0 | 0 | 1
Pyelonephritis (Infections and infestations) | 0 | 0 | 1
Skin infection (Infections and infestations) | 1 | 0 | 0
Soft tissue infection (Infections and infestations) | 0 | 1 | 0
Streptococcal bacteraemia (Infections and infestations) | 1 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 1 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 3 | 0 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Procedural haemorrhage (Injury, poisoning and procedural complications) | 0 | 1 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 1 | 0 | 0
Neutrophil count decreased (Investigations) | 1 | 1 | 1
Blood bilirubin increased (Investigations) | 0 | 1 | 1
Ejection fraction decreased (Investigations) | 0 | 1 | 0
Liver function test increased (Investigations) | 1 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hypovolaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Pathological fracture (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Spinal pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Encephalopathy (Nervous system disorders) | 0 | 1 | 0
Haemorrhage intracranial (Nervous system disorders) | 0 | 1 | 0
Headache (Nervous system disorders) | 0 | 1 | 0
Loss of consciousness (Nervous system disorders) | 1 | 0 | 0
Seizure (Nervous system disorders) | 0 | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 1 | 0
Hydronephrosis (Renal and urinary disorders) | 0 | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 4 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pneumothorax spontaneous (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Embolism (Vascular disorders) | 0 | 1 | 0
Haematoma (Vascular disorders) | 1 | 0 | 0
Subclavian vein thrombosis (Vascular disorders) | 1 | 0 | 0
Vasculitis (Vascular disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Margetuximab Plus Chemotherapy (N=264) | Trastuzumab Plus Chemotherapy (N=266) | Margetuximab Infusion Substudy (N=88)
Neutropenia (Blood and lymphatic system disorders) | 72 | 54 | 17
Anaemia (Blood and lymphatic system disorders) | 48 | 61 | 18
Thrombocytopenia (Blood and lymphatic system disorders) | 22 | 13 | 3
Nausea (Gastrointestinal disorders) | 88 | 87 | 33
Diarrhoea (Gastrointestinal disorders) | 68 | 67 | 14
Constipation (Gastrointestinal disorders) | 50 | 44 | 20
Vomiting (Gastrointestinal disorders) | 55 | 38 | 19
Abdominal pain (Gastrointestinal disorders) | 25 | 36 | 9
Stomatitis (Gastrointestinal disorders) | 28 | 21 | 8
Abdominal pain upper (Gastrointestinal disorders) | 22 | 21 | 1
Dyspepsia (Gastrointestinal disorders) | 16 | 20 | 7
Fatigue (General disorders) | 112 | 95 | 24
Pyrexia (General disorders) | 50 | 34 | 18
Asthenia (General disorders) | 49 | 32 | 7
Oedema peripheral (General disorders) | 21 | 26 | 5
Mucosal inflammation (General disorders) | 26 | 8 | 3
Influenza like illness (General disorders) | 18 | 11 | 5
Urinary tract infection (Infections and infestations) | 25 | 26 | 5
Upper respiratory tract infection (Infections and infestations) | 21 | 23 | 7
Nasopharyngitis (Infections and infestations) | 21 | 19 | 1
Infusion related reaction (Injury, poisoning and procedural complications) | 33 | 9 | 18
Neutrophil count decreased (Investigations) | 32 | 38 | 12
Aspartate aminotransferase increased (Investigations) | 22 | 34 | 12
Alanine aminotransferase increased (Investigations) | 26 | 26 | 11
White blood cell count decreased (Investigations) | 20 | 26 | 8
Weight decreased (Investigations) | 16 | 15 | 9
Decreased appetite (Metabolism and nutrition disorders) | 38 | 38 | 9
Hypokalaemia (Metabolism and nutrition disorders) | 16 | 21 | 8
Pain in extremity (Musculoskeletal and connective tissue disorders) | 32 | 25 | 7
Arthralgia (Musculoskeletal and connective tissue disorders) | 28 | 23 | 10
Back pain (Musculoskeletal and connective tissue disorders) | 23 | 27 | 7
Myalgia (Musculoskeletal and connective tissue disorders) | 18 | 16 | 4
Muscle spasms (Musculoskeletal and connective tissue disorders) | 17 | 11 | 7
Headache (Nervous system disorders) | 50 | 43 | 11
Neuropathy peripheral (Nervous system disorders) | 26 | 28 | 7
Dizziness (Nervous system disorders) | 26 | 17 | 5
Dysgeusia (Nervous system disorders) | 16 | 15 | 7
Peripheral sensory neuropathy (Nervous system disorders) | 17 | 13 | 3
Insomnia (Psychiatric disorders) | 15 | 15 | 6
Cough (Respiratory, thoracic and mediastinal disorders) | 42 | 33 | 6
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 34 | 29 | 13
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 18 | 19 | 2
Alopecia (Skin and subcutaneous tissue disorders) | 47 | 39 | 13
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 33 | 43 | 1
Rash (Skin and subcutaneous tissue disorders) | 18 | 15 | 6
Pruritus (Skin and subcutaneous tissue disorders) | 13 | 13 | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2020-06-08): https://cdn.clinicaltrials.gov/large-docs/11/NCT02492711/Prot_000.pdf
  • Statistical Analysis Plan (2018-03-13): https://cdn.clinicaltrials.gov/large-docs/11/NCT02492711/SAP_001.pdf